CLINICAL TRIAL: NCT06548516
Title: Evaluation of Patients' Perceptions and Soft Tissue Changes After Conventional and Diode Laser Frenectomy
Brief Title: Maxillary Labial Frenectomy: Diode Lasers Versus Surgical Scalpel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeynep Tastan Eroglu, Assistant professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: frenektomilaserandconvantional
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: High Frenum Attachment
Keywords: Maxillary Labial Frenum; Frenectomy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Masking Description: Patients in the C group underwent primary wound healing with sutures, whereas patients in the L group did not get any sutures. Therefore, neither the clinicians (Z.T.E and K.Y) nor the patients were kept unaware of the study's details over the entire duration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (conventional scalpel surgery) (Active Comparator): After administering local infiltrative anesthesia with articaine hydrochloric acid combined with epinephrine 1:100,000, the frenum will be grasped with a straight hemostat positioned in the vestibule. The tissue adjacent to the upper and lower surfaces of the hemostat will then be incised using a no.15 scalpel. The excised diamond-shaped portion of the frenum will be removed with the hemostat. Subsequently, a horizontal incision will be made on the periosteum with a scalpel to prevent fiber reattachment. The wound site will be primarily closed using absorbable sutures (4/0, Pegelak), which will be removed one week post-operatively.
  Interventions: Procedure: Control group (conventional scalpel surgery)
- Diode laser group (Experimental): The frenectomy procedure will be performed under local infiltrative anesthesia, specifically articaine hydrochloric acid with epinephrine 1:100,000. A straight hemostat, similar to that used in the C group, will be employed to secure the frenum. Laser energy will be applied to the upper and lower sections of the frenum adjacent to the hemostat, utilizing a diode laser device equipped with a 400 µm diameter, plain-ended optical fiber tip. Frenectomy will performed with a 980 nm diode laser with 1.7 W power in continuous wave mode.The wound site will be allowed to heal by secondary intention without the application of sutures.
  Interventions: Procedure: Diode laser group

INTERVENTIONS:
Procedure: Control group (conventional scalpel surgery) — The patients in the control group will undergo frenectomy using conventional scalpel surgery.
  Arms: Control group (conventional scalpel surgery)
Procedure: Diode laser group — The patients in the laser group will undergo frenectomy using a diode laser.
  Arms: Diode laser group

SUMMARY:
The goal of this clinical trial is to determine if diode laser treatment can improve post-operative outcomes compared to conventional scalpel technique in systemically healthy, non-smoking adults aged 18-45 years with aberrant papillary frenum attachment. The main questions it aims to answer are:

Does diode laser treatment result in lower post-operative pain compared to the conventional scalpel technique? Does diode laser treatment result in better periodontal healing outcomes compared to the conventional scalpel technique? Researchers will compare the diode laser surgery group to the conventional scalpel surgery group to see if there are differences in pain and healing.

Participants will:

Undergo a frenectomy procedure using either a diode laser or a conventional scalpel.

Receive oral hygiene instructions and post-operative care recommendations. Have their periodontal parameters measured at baseline, 6 weeks, and 6 months post-operation.

Record their pain levels using a visual analogue scale on specified post-operative days.

DETAILED DESCRIPTION:
The trial will be performed as a prospective, randomized and controlled, single-blind investigation to study clinical parameters and patients' experiences when performing a frenectomy, comparing diode laser treatment with the conventional scalpel technique.

Participants:

This study will include 43 participants who will be identified with aberrant papillary frenum attachment according to Mirko et al., and will be referred to the periodontology department. The inclusion criteria for the participants will be:

All participants will sign a written informed consent form before participating in the study.

Study Groups and Randomization:

Before any surgical procedure, all subjects will undergo a thorough medical and dental history review, as well as intraoral and radiographic examinations. Participants who match the inclusion criteria will be provided with oral hygiene instructions tailored to their specific needs. Initially, the clinical periodontal parameters of all participants will be measured. Then, a mechanical cleaning procedure will be carried out using an ultrasonic scaler (CavitronÒ; Dentsply International) and hand instruments (Gracey, 5/6, 7/8, 11/12, 13/14; Hu-Friedy Ins. Co.). A total of 43 participants will be enrolled in the study and assigned to one of two groups using a computer-based randomization table (www.graphpad.com/quickcalcs). The participants will be randomly divided into two groups: the experimental group, which will undergo diode laser surgery (L=20), and the control group, which will undergo conventional scalpel surgery (C=23).

Post-treatment Procedure:

After the frenectomy procedures in all groups, patients will receive oral hygiene instructions and will be advised to consume soft and cold food for the next 12 hours. Additionally, a 0.12% chlorhexidine gluconate mouth rinse will be prescribed to be used once a day for one minute over five days. For pain relief, 500 mg of acetaminophen (1-2 tablets) will be prescribed as needed, with patients instructed to record the dosage and frequency of use.

Clinical Evaluation:

Z.T.E. will perform all surgical procedures, while a calibrated single examiner (K.Y) will perform all clinical evaluations. Patients in the C group will undergo primary wound healing with sutures, whereas patients in the L group will not get any sutures. Therefore, neither the clinicians (Z.T.E and K.Y) nor the patients will be kept unaware of the study's details over the entire duration. In order to ensure consistency in the measurements of K.Y, a calibration exercise was conducted until the agreement coefficient achieves a level of 90%. This calibration process was consist of evaluating three patients on two separate occasions within a 24-hour period. The calibration was considered effective if the variation between repeated measurements of periodontal keratinized gingival width (KGW) at the beginning and after 24 hours is less than 3%. The clinical periodontal parameters, such as the plaque index (PI), gingival index (GI), and periodontal pocket depth (PD), will be measured using a periodontal probe from the University of North Carolina (PCPUNC15; Hu-Friedy Ins. Co.). At baseline and at postoperative week 6 and month 6, all periodontal measurements will be taken at six sites per tooth as part of a full-mouth evaluation. KGW on teeth 11 and 12, the heights of the interdental papillae between the incisors (from the tip of an interdental papilla to the line joining the lowest points on the gingival margins of adjacent incisors), interdental papilla width, and the amount of diastema will be measured at baseline and at month 6. Before the operations, the labial frenulum attachments will be classified into four types: I - mucosal attachment; II - gingival attachment; III - papillary attachment; and IV - papilla penetrating attachment. Pain will be evaluated using the visual analogue scale (VAS) on postoperative days 1, 3, 7, 14, 21, and 28. The scale will be comprised of a horizontal line with values ranging from '0' to '10', where '0' indicates the absence of pain and '10' indicates the presence of severe discomfort.

Statistical Analysis:

Each patient will be accepted as one statistical unit and the statistical analysis will be performed by SPSS 20 (SPSS Corporation, Chicago, IL) with a significance level p < 0.05. The Kolmogorov-Smirnov test will be used to check the distribution for normality. Repeated measurements of clinical parameters will be analyzed with Friedman test and Wilcoxon signed-rank test. The Kruskal-Wallis, Chi-square, and Fisher's exact tests will be used to determine differences among the groups. Moreover, in case of significant difference among groups, the Mann-Whitney U test will be used to compare two groups by Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Nonsmoker
* No periodontal treatment received in the last 3 months
* Having at least 20 teeth
* Presence of at least central incisors, lateral incisors, and canines in the maxilla
* Not pregnant or breastfeeding
* No psychiatric, mental, or physical impairments
* Diagnosed with gingival health based on the "World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions
* Consent to participate in the study.

Exclusion Criteria:

* Any systemic disease that could interfere with the wound healing process (e.g., diabetes mellitus and HIV infection)
* Smoking
* Use of antibiotics, anti-inflammatory drugs, or any other medication in the last 6 months that could affect the study's outcome
* Any hypersensitivity reactions to paracetamol
* Any physical limitations or restrictions that could impede normal oral hygiene procedures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | postoperative days 1, 3, 7, 14, 21, and 28.
  Pain will be evaluated using the visual analogue scale (VAS).The scale will be comprised of a horizontal line with values ranging from '0' to '10', where '0' indicates the absence of pain and '10' indicates the presence of severe discomfort.
Postoperative tissue healing | postoperative days 7 and 30 after surgery,
  Tissue healing will be assessed by Z.T.E using the following scoring system:
  * Score 1: Complete epithelialization
  * Score 2: Incomplete epithelialization
  * Score 3: Presence of ulcer
  * Score 4: Tissue defect or necrosis

CONTACTS AND LOCATIONS:
Overall Officials: zeynep taştan eroğlu, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, dentistry Faculty, Konya, Turkey (Türkiye)